CLINICAL TRIAL: NCT01417598
Title: Improving Balance Function in Elderly by Progressive and Specific Training and Physical Activity- a Randomized Controlled Study.
Brief Title: BETA Study: Improving Balance Function in Elderly by Progressive and Specific Training and Physical Activity
Acronym: BETA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Alexandra Halvarsson, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K2011-69P-20908-02-4
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Elderly; Parkinsons Disease; Osteoporosis
Keywords: Balance; Gait; Physical activity
MeSH Terms: conditions — Parkinson Disease; Osteoporosis; Motor Activity | interventions — Gait; Nordic Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gait and balance group training (Experimental): The balance-training program is based on scientifically well-established principles of exercise training and postural control as well as current research on training in elderly and PD. For the PD group it has been modified based on the current knowledge of the neurophysiology and the inevitable constraints on mobility and postural control resulting from basal ganglia degeneration. The training will be conducted as a progressive individually adjusted group program, led by experienced physiotherapists and researchers in order to challenge the specific balance disorder of every participant and endorse progression. It is progressive and specific balance program including dual- and multitasks. The program is performed 3 times/week for 10-12 weeks.
  Interventions: Other: Gait and balance group training
- Gait and balance trainig + nordic walking (Experimental): (only for Osteoporosis group)
  Interventions: Other: Nordic walking (only osteoporosis group)
- Control group (No Intervention)

INTERVENTIONS:
Other: Gait and balance group training — The balance-training program is based on scientifically well-established principles of exercise training and postural control as well as current research on training in elderly and PD. For the PD group it has been modified based on the current knowledge of the neurophysiology and the inevitable constraints on mobility and postural control resulting from basal ganglia degeneration. The training will be conducted as a progressive individually adjusted group program, led by experienced physiotherapists and researchers in order to challenge the specific balance disorder of every participant and endorse progression. It is progressive and specific balance program including dual- and multitasks. The program is performed 3 times/week for 10-12 weeks.
  Arms: Gait and balance group training
Other: Nordic walking (only osteoporosis group) — To further test the hypothesis that physical activity may enhance the results from the balance training program pole striding will be added to the balance training program, at least 30-45 minutes three times per week during leisure time. Each individual in this group will be provided with individually adjusted poles, a pedometer and a diary to enter when and for how long time they have been walking.
  Arms: Gait and balance trainig + nordic walking

SUMMARY:
Balance control, physical activity and health related quality of life will be assessed before and after a 10 to 12 weeks training program as well as 6 and 12 months thereafter in 200 elderly (>60) with balance problems (100 with osteoporosis, 100 with Parkinson's disease). Osteoporosis subjects will be assigned to 3 groups (balance training, balance training and Nordic walking, or control group) and Parkinson's subjects to 2 groups (balance training or a control group). The training will be progressive and specific incorporating dual task exercises (directly related to an increased risk of falling). Clinical and laboratory gait and balance measures as well as questionnaires will be used to assess physical function and quality of life. An earlier study, investigating this training program in healthy elderly with balance problems showed that the training was well-tolerated and effective, with a significant increase in balance control, physical function and activity. In this study, we expect that an improvement in balance function, physical activity and health related quality of life, which will lead to a decreased number of falls, prevent and/or postpone incidence of a hazardous fall and thereby reduce the burden on the health care system. Our model for functional balance training and outcome methods will expand techniques and tools available to physical therapists and health care scientist treating and evaluating patients with loss of balance function. Elderly receiving therapy with the goal to improve or recuperate physical function and balance will benefit from this project.

ELIGIBILITY:
* Osteoporosis: To be included the candidate must: be >65 years with osteoporosis objectively verified by Dual energy X-ray absorptiometry (DXA) in the hip and lumbar back,be an independent ambulator, have experienced at least one fall in the last 12 months and have an adequate medical treatment for their osteoporosis.
* Parkinson's disease: All PD subjects will have a clinical diagnosis of -idiopathic‖ PD (Hoehn &Yahr scores 2-3), > 60 years of age and no other existing neuromuscular disorders, including severely flexed posture. In addition, the subjects will have no history suggesting -atypical‖ PD symptoms.

Exclusion criteria's for all subjects are:

* moderate-severe dementia (Mini-Mental score <24)
* respiratory, cardiovascular, musculoskeletal or neurological (except PD) disorders that may interfere with participation in the exercise program

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2016-06 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Improved balance control | Short-term
Improved gait | Short-term
Improved physical activity | Long-term
Reduced Fear of falling | Short-term

SECONDARY OUTCOMES:
Improved health related quality of life | Long-term

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Huddinge, Sweden

REFERENCES:
- [Derived] Rennie L, Opheim A, Dietrichs E, Lofgren N, Franzen E. Highly challenging balance and gait training for individuals with Parkinson's disease improves pace, rhythm and variability domains of gait - A secondary analysis from a randomized controlled trial. Clin Rehabil. 2021 Feb;35(2):200-212. doi: 10.1177/0269215520956503. Epub 2020 Sep 28. PMID 32985265
- [Derived] Lofgren N, Conradsson D, Joseph C, Leavy B, Hagstromer M, Franzen E. Factors Associated With Responsiveness to Gait and Balance Training in People With Parkinson Disease. J Neurol Phys Ther. 2019 Jan;43(1):42-49. doi: 10.1097/NPT.0000000000000246. PMID 30531385
- [Derived] Lofgren N, Conradsson D, Rennie L, Moe-Nilssen R, Franzen E. The effects of integrated single- and dual-task training on automaticity and attention allocation in Parkinson's disease: A secondary analysis from a randomized trial. Neuropsychology. 2019 Feb;33(2):147-156. doi: 10.1037/neu0000496. Epub 2018 Nov 8. PMID 30407031
- [Derived] Conradsson D, Nero H, Lofgren N, Hagstromer M, Franzen E. Monitoring training activity during gait-related balance exercise in individuals with Parkinson's disease: a proof-of-concept-study. BMC Neurol. 2017 Jan 31;17(1):19. doi: 10.1186/s12883-017-0804-7. PMID 28143463
- [Derived] Conradsson D, Lofgren N, Stahle A, Hagstromer M, Franzen E. A novel conceptual framework for balance training in Parkinson's disease-study protocol for a randomised controlled trial. BMC Neurol. 2012 Sep 27;12:111. doi: 10.1186/1471-2377-12-111. PMID 23017069